CLINICAL TRIAL: NCT04579406
Title: Association of Changes in NPY, CGRP, SP and TRPV1 With Perioperative Adverse Cardiovascular Event in Type-2 Diabetic Patients
Brief Title: Perioperative Adverse Cardiovascular Event in Type-2 Diabetic Patients
Acronym: DMPACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, Professor and chairman of the Department of Anesthesiology, Second Hospital of Shanxi Medical University
Other Study IDs: ScondShanxiMU-1646
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes; Neuropathy
Keywords: Diabetes mellitus; adverse cardiovascular events; nerve degeneration; peripheral sensory nerves
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Nerve Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-diabetic group: The non-diabetic patients undergoing non-cardiac surgery.
  Interventions: Procedure: non-cardiac surgery
- Diabetic group: The diabetic patients without peripheral neuropathy undergoing non-cardiac surgery.
  Interventions: Procedure: non-cardiac surgery
- Diabetic neuropathic group: The diabetic patients with peripheral neuropathy undergoing non-cardiac surgery.
  Interventions: Procedure: non-cardiac surgery

INTERVENTIONS:
Procedure: non-cardiac surgery — All the patients are undergoing non-cardiac surgery.

SUMMARY:
The study was designed to investigate the correlation between perioperative adverse cardiovascular events and the degeneration of sensory nerves in patient diagnosed with type 2 diabetes mellitus, undergoing elective non-cardiac surgery.

DETAILED DESCRIPTION:
The study was designed to investigate the correlation between perioperative adverse cardiovascular events and the degeneration of sensory nerves in patient diagnosed with type 2 diabetes mellitus, undergoing elective non-cardiac surgery. Diabetes mellitus and peripheral sensory nerve degeneration will be diagnosed via clinical evaluation. Serum levels of constituent neuropeptides, including neuropeptide Y (NPY), calcitonin and substance P (SP) and calcitonin gene related peptide (CGRP), and transient receptor potential vanilloid 1 (TRPV1), a molecular nociceptor in peripheral sensory nerves will be quantitatively evaluated. The clinical and the biochemical consequence will be compared between the cohorts of diabetic and non-diabetic patients. The differences and the correlations will be analyzed. The results of the study may reveal whether or not the perioperative adverse cardiovascular events in diabetic patients are correlated with degeneration of peripheral sensory nerves and the alterations in the neuropeptides and TRPV1 are potentially applicable for evaluation of the risk of cardiovascular events in perioperative period in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* The main discharge diagnosis is T2DM；
* Age > 18 years old;
* No acute complications of diabetes

Exclusion Criteria:

* T1DM patients;
* EGFR < 60 ml/min/1.73 m or proteinuria (or both);
* Patients with history of acute cardiovascular events;
* Familial hypercholesterolemia or other hereditary lipid metabolism diseases;
* anti-HIV patients;
* Patients with serious mental health problems;
* Patients receiving drugs that can lead to dyslipidemia, such as antipsychotics, corticosteroids, or immunosuppressants;
* Patients with systemic inflammatory diseases, such as systemic lupus erythematosus;
* Patient are quitting smoking and severe obesity (BMI>40)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic patients with and without peripheral sensory neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
adverse cardiovascular events | Perioperative period
  All the pre-, intra- and post-operative adverse cardiovascular events in the patients will be taken into account.

SECONDARY OUTCOMES:
NPY, CGRP, SP and TRPV1 | Perioperative period
  The difference in the serum levels of NPY, CGRP, SP and TRPV1

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Guo, M.B., Ph.D., Study Director — Second Hospital of Shanxi Medical University
Locations (1):
- Zheng Guo, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided
Yes, if possible.